CLINICAL TRIAL: NCT05058924
Title: Low Molecular Weight hEparin vs. Aspirin Post-partum
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0275A
Record Dates: First submitted 2021-08-25; First posted 2021-09-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism
Keywords: Postpartum; Prophylaxis; LMWH
MeSH Terms: conditions — Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight; Aspirin

STUDY DESIGN:
Intervention Model Description: Single Center pilot feasibility RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Low Molecular Weight Heparin (LMWH) (Active Comparator): Prophylactic LMWH for 6 weeks postpartum
  Interventions: Drug: Prophylactic low molecular weight heparin
- Prophylactic Low Molecular Weight Heparin (LMWH) + Low Dose Aspirin (Experimental): Prophylactic LMWH for 3 weeks followed by low dose Aspirin for 3 weeks.
  Interventions: Drug: Low molecular weight heparin and low-dose aspirin

INTERVENTIONS:
Drug: Prophylactic low molecular weight heparin — Enoxaparin 40 mg/dalteparin 5000 U/tinzaparin 4500 U subcutaneously daily for women with weight <100 kg for 6 weeks.
  Other Names: LMWH
  Arms: Prophylactic Low Molecular Weight Heparin (LMWH)
Drug: Low molecular weight heparin and low-dose aspirin — Enoxaparin 40 mg/dalteparin 5000 U/tinzaparin 4500 U subcutaneously daily for women with weight <100 kg for three weeks followed by ASA 81 mg orally daily for three weeks.
  Other Names: LMWH; ASA
  Arms: Prophylactic Low Molecular Weight Heparin (LMWH) + Low Dose Aspirin

SUMMARY:
This is single centre pilot, randomized controlled trial assessing postpartum prophylactic anticoagulation with 3 weeks of LMWH followed by 3 weeks of Aspirin compared to standard of care of prophylactic LMWH for 6 weeks at moderate to high risk of developing VTE.

DETAILED DESCRIPTION:
A single centre pilot, randomized controlled trial assessing postpartum prophylactic anticoagulation with 3 weeks of LMWH followed by 3 weeks of Aspirin compared to standard of care of prophylactic LMWH for 6 weeks for women at moderate to high risk of developing VTE to determine feasibility of conducting a large non inferiority trial using the same regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Personal history of unprovoked VTE prior to pregnancy or hormone associated VTE and not prescribed therapeutic anticoagulation or
2. Family history (1st degree relative) of VTE and antithrombin deficiency, protein C or protein S deficiency or
3. Combined thrombophilia or homozygous for the factor V Leiden mutation or prothrombin gene mutation, and family history of VTE (1st degree relative) and
4. > 18 years of age.

Exclusion Criteria:

1. Pre-existing indication for therapeutic LMWH
2. Contraindication to ASA:

   1. Known ASA allergy
   2. Documented history of gastrointestinal ulcer
   3. Known platelet count < 50x10^9/L at any time during the current pregnancy or postpartum
3. Contraindication to LMWH, e.g. known allergy
4. Active bleeding at any site, excluding physiological vaginal bleeding
5. Patients with bleeding disorders
6. Known severe hypertension (SBP >200mm/hg and/or DBP >120mm/hg) during the current pregnancy or postpartum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | 1 year
Consent Rate | 1 year
Adherence to Prescription | 6 weeks
  Utilization of co-interventions for both: control group (6 week of Low Molecular Weight Heparin) or Treatment group (3 week of low molecular weight Heparin and 3 week of low dose aspirin).
Withdrawal of consent rate | 1 year
Rates of contamination | 6 weeks
  List of the concurrent medication will be gathered on 3 week follow up, 6 week follow up and early discontinuation (before 6 weeks).

SECONDARY OUTCOMES:
VTE event rate | 3 months
  VTE must be confirmed either by Doppler ultrasound or V/Q scan or computer tomography (CT). Imaging will not be performed on all patients, only those with symptoms of VTE event. Event rate of VTE will be calculated by number of VTE events by Total days in this study. This number of VTE event is collected during 3 week follow up, 6 week follow up, 3 months follow-up and on early discontinuation date (before 3 months follow up). At the end of the study (after 3 month), the total VTE event rate is calculated.
Bleeding assessment six weeks following delivery | 6 weeks
  According to the International Society on Thrombosis and Hemostasis (ISTH) scoring system. The bleeding assessments are collected on 3 week phone call and 6 week phone call or early discontinuation visit (before 6 week follow up)
Anticoagulation Satisfaction Assessment using the PACT Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Shehata, MD, Principal Investigator — Department of Medicine/IHPME, University of Toronto, Division of Hematology, Mount Sinai Hospital; Evanglia Vlachodimitropoulou Koumoutsea, MBBS, Principal Investigator — Department of Obstetrics and Gynecology, University of Toronto, Mount Sinai Hospital
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matharu GS, Kunutsor SK, Judge A, Blom AW, Whitehouse MR. Clinical Effectiveness and Safety of Aspirin for Venous Thromboembolism Prophylaxis After Total Hip and Knee Replacement: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Intern Med. 2020 Mar 1;180(3):376-384. doi: 10.1001/jamainternmed.2019.6108. PMID 32011647
- [Background] Bates SM, Rajasekhar A, Middeldorp S, McLintock C, Rodger MA, James AH, Vazquez SR, Greer IA, Riva JJ, Bhatt M, Schwab N, Barrett D, LaHaye A, Rochwerg B. American Society of Hematology 2018 guidelines for management of venous thromboembolism: venous thromboembolism in the context of pregnancy. Blood Adv. 2018 Nov 27;2(22):3317-3359. doi: 10.1182/bloodadvances.2018024802. PMID 30482767
- [Result] Samsa G, Matchar DB, Dolor RJ, Wiklund I, Hedner E, Wygant G, Hauch O, Marple CB, Edwards R. A new instrument for measuring anticoagulation-related quality of life: development and preliminary validation. Health Qual Life Outcomes. 2004 May 6;2:22. doi: 10.1186/1477-7525-2-22. PMID 15132746
- [Result] Rodeghiero F, Tosetto A, Abshire T, Arnold DM, Coller B, James P, Neunert C, Lillicrap D; ISTH/SSC joint VWF and Perinatal/Pediatric Hemostasis Subcommittees Working Group. ISTH/SSC bleeding assessment tool: a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders. J Thromb Haemost. 2010 Sep;8(9):2063-5. doi: 10.1111/j.1538-7836.2010.03975.x. No abstract available. PMID 20626619
- [Result] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Result] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Derived] Vlachodimitropoulou E, Malinowski K, Kaplovitch E, Carrier M, Shehata N. Low-molecular-weight heparin vs aspirin postpartum (LEAP): a single-center pilot randomized control trial. Blood Vessel Thromb Hemost. 2025 Sep 10;2(4):100106. doi: 10.1016/j.bvth.2025.100106. eCollection 2025 Nov. PMID 41280308

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05058924/Prot_004.pdf
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT05058924/ICF_006.pdf